CLINICAL TRIAL: NCT01561573
Title: Ultrasound Assisted Distal Radius Fracture Reduction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Andrew Skinner, Dr. William Andrew Skinner, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPH-POCUS-2012
Record Dates: First submitted 2012-03-16; First posted 2012-03-23 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Colles Fracture; Point of Care Ultrasound; Emergency Ultrasound
Keywords: Point of Care Ultrasound; Emergency Ultrasound; Colles Fracture; Fracture Reduction; Bedside Ultrasound
MeSH Terms: conditions — Colles' Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound colles fracture (Other): This is a single arm study
  Interventions: Device: Point of care ultrasound

INTERVENTIONS:
Device: Point of care ultrasound — A bedside ultrasound machine will be used to image the colles fracture during the fracture reduction process.
  Other Names: Ultrasound Machines used in the study will include; Sonosite micromaxx; Sonosite M-Turbo; Ultrasonix Sonixtouch; Ultrasonix Sonixtablet; Esaote MyLab Five; Esaote MyLab 25 Gold

SUMMARY:
PURPOSE: to evaluate the utility of bedside ultrasound performed by emergency physicians in the evaluation and reduction of colles fractures as compared with traditional pre and post reduction radiographs. With the objectives of assessing Emergency Ultrasounds (EU) utility in guiding reduction attempts of Colles fractures and to compare EU to x-ray for the final assessment of reduction adequacy.

DETAILED DESCRIPTION:
The reduction of fractures is a commonly performed procedure in emergency departments (EDs). In most Canadian EDs, reductions are performed by emergency physicians (EPs). The distal radius fracture is the most common fracture requiring reduction. Fracture reduction is time-consuming with several steps required: initial evaluation including x-ray, equipment and personnel gathering, sedation and/or local anesthesia, reduction attempt(s) and splinting/casting, and post-reduction x-rays, with subsequent patient reassessment. These steps have a negative effect on ED patient throughput. Subsequent to the reduction attempt(s), the patient is sent for x-ray often with uncertainty regarding the reduction success. Fluoroscopy is generally not an option for the EP in evaluating accuracy of reduction. If the reduction is not adequate, further reduction attempts are needed. This utilizes more resources, either in the ED or orthopedic clinic or operating room, depending on where further reduction attempts are made.

Emergency ultrasound (EU) in Canada has become a well-established part of emergency medical practice in recent years as evidenced by the latest position statement of the Canadian Association of Emergency Physicians (http://caep.ca/template.asp?id=B5283F4158FB471AA56E480D6277C1AC) and the development of the Canadian Emergency Ultrasound Society (www.ceus.ca). A growing body of literature has shown the utility of EU in the diagnosis and reduction of fractures (1-6). A recent case report (7) showed that EU can be used to aid Colles fracture reduction. Similar to fluoroscopy, EU may be a fast and accurate method of determining successful fracture reduction. Unlike fluoroscopy, EU is available immediately in the ED. EU may also obviate the need for the post-reduction x-ray, particularly in the setting where the patient will have yet another x-ray at the time of orthopedic follow-up to evaluate for interval loss of reduction. Thus, EU has the potential to significantly reduce time to discharge.

Our study has the following objectives:

* To assess EU utility for guiding reduction attempts of distal radius fractures.
* To compare EU to x-ray for the final assessment of reduction adequacy.

ELIGIBILITY:
Inclusion Criteria:

* > 19 years old
* Able to provide voluntary and informed consent
* Distal radius fracture is the main traumatic injury
* Planned reduction to be performed by the EP
* Treating EP trained to perform EU for fractures OR one of the study authors available to perform EU

Exclusion Criteria:

* < 19 years old
* Patient unable to provide voluntary and informed consent
* Distal radius fracture is only one of several significant injuries
* No reduction to be performed by the EP
* EP not trained to perform EU for fractures AND no study author available to perform EU

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Point of care ultrasound in Identifying colles fracture reduction | 1 year
  Physicians performing Bedside ultrasound of colles fractures will be asked to complete likert scales on the adequacy of fracture reduction with ultrasound

SECONDARY OUTCOMES:
Number of reduction attempts affected by ultrasound | 1 year
  The physician is asked to record the number of fracture reduction attempts as guided by the ultrasound image before and after the post reduction X-ray
Time to imaging | 1 year
  The physician performing the bedside ultrasound will record the time on completion of the bedside ultrasound and the time of completion of the post reduction X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Skinner, MD, Principal Investigator — St. Paul's Hospital; Steve Socransky, MD, Study Director — Sudbury Regional Hospital; Ray Wiss, MD, Study Director — Sudbury Regional Hospital
Locations (8):
- Canada (8):
  - Foothills Medical Center, Calgary, Alberta
  - Namnaimo General Hospital, Nanaimo, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - St. John's Health Science Center, St. John's, Newfoundland and Labrador
  - Dartmouth General Hospital, Dartmouth, Nova Scotia
  - Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Toronto East General Hospital, Toronto, Ontario